CLINICAL TRIAL: NCT02413606
Title: ENdometrial Cancer SURvivors' Follow-up carE (ENSURE): Less is More? Randomized Controlled Trial to Evaluate Patient Satisfaction and Cost-effectiveness of a Reduced Follow-up Schedule
Brief Title: ENdometrial Cancer SURvivors' Follow-up carE (ENSURE): Less is More?
Acronym: ENSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comprehensive Cancer Centre The Netherlands (Other)
Collaborators: Dutch Cancer Society (Other); Maastricht University Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Nicole Ezendam, Dr., Comprehensive Cancer Centre The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IKZ 2014-6677
Record Dates: First submitted 2015-03-24; First posted 2015-04-10 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Cancer
Keywords: follow up care; satisfaction with care
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): reduced follow-up schedule: 4 follow-up visits, after 3, 12, 24 and 36 months
  Interventions: Other: Reduced follow-up schedule
- control (No Intervention): regular follow-up schedule according to the guideline, 10-13 visits during 5 years

INTERVENTIONS:
Other: Reduced follow-up schedule — In the intervention group, the follow-up schedule will be limited to four follow-up visits at 3, 12, 24 and 36 months, under the specific condition that patients have easy and prompt access to care (specialised nurse of gynaecologist) if symptoms or questions occur. The content of the follow-up visits will be similar for both groups.
  Arms: Intervention

SUMMARY:
Background: It has often been hypothesized that the frequency of follow-up for patients with early-stage endometrial cancer could be decreased. However, studies evaluating effects of a reduced follow-up schedule among this patient group are lacking.

Objective: Assess patient satisfaction and cost-effectiveness of a less frequent follow-up schedule compared to the schedule according to the Dutch guideline.

Study design: Dutch multicentre randomized controlled trial with a 5 year follow-up. Patients (n=282) are randomized in an intervention group with 4 follow-up visits during 3 years, and a control group with 10-13 follow-up visits during 5 years, according to the Dutch guideline. Patients are asked to fill out a questionnaire at baseline, 6, 12, 36 and 60 months. Patient inclusion will take two years (if 60% of the patients participate).

Outcomes: Primary: Patient satisfaction with follow-up care and cost-effectiveness.

Secondary: health care use, adherence to schedule, health-related quality of life, fear of recurrence, anxiety and depression, information provision, recurrence, survival

Patients: Stage 1A and 1B low-risk endometrial cancer patients, for whom adjuvant radiotherapy is not indicated

Statistics: linear regression analyses to assess differences in patient satisfaction with follow-up care between intervention and control group adjusted for potential pre-defined confounders.

Expected results: Patients in the intervention arm have a similar satisfaction with follow-up care and overall outcomes, but lower health care use and costs than patients in the control arm. No effects are expected on QALY differences (losses) and satisfaction, but the reduced schedule is expected to save 144.000 per year in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Endometrioïd type endometrial carcinoma with stage 1 (FIGO, 2009) disease, with the following combination of stage, age and grade:

   Stage 1A, any age, grade 1 or 2; Stage 1B, < 60 years, grade 1 or 2 without LVSI;
2. Written informed consent;
3. Sufficient oral and written command of the Dutch language.

Exclusion Criteria:

1. Any other stage and type of endometrial carcinoma
2. Histological types papillary serous carcinoma or clear cell carcinoma
3. Uterine sarcoma (including carcinosarcoma)
4. Radiotherapy for current endometrial carcinoma
5. Previous malignancy (except for non-melanomatous skin cancer) < 5 yrs
6. Confirmed Lynch syndrome
7. Previous pelvic radiotherapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with follow-up care | up to 60 months after completion of primary treatment
  assessed with the PSQIII questionnaire; analysed with a repeated mixed model as one overall outcome over all time points
Costs-effectiveness | assessed at 60 months after completion of primary treatment
  Cost-effectiveness from the health care perspective using the EQ-5D

SECONDARY OUTCOMES:
Costs-effectiveness | assessed at 36 months after completion of primary treatment
  Cost-effectiveness from the health care perspective using the EQ-5D
Health care use -gynaecologist, (specialist) nurse, primary care physician and other health or care services-; adherence to the indicated follow-up protocols; reasons for non-adherence | assessed at 6, 12 and 36 months after completion of primary treatment
  health care use is assessed from hospital charges, primary care physician and self-report; analysed with a repeated mixed model as one overall outcome over all time points
Health care use -gynaecologist, (specialist) nurse, primary care physician and other health or care services-; adherence to the indicated follow-up protocols; reasons for non-adherence | assessed at 6, 12, 36, and 60 months after completion of primary treatment
  health care use is assessed from hospital charges, primary care physician and self-report; analysed with a repeated mixed model as one overall outcome over all time points
Health-Related Quality of Live | assessed at baseline, 6, 12, and 36 months after completion of primary treatment
  assessed with questionnaires: EORTC QLQ-C30 and EORTC QLQ-EN24; analysed with a repeated mixed model as one overall outcome over all time points
Health-Related Quality of Live | assessed at baseline, 6, 12, 36, and 60 months after completion of primary treatment
  assessed with questionnaires: EORTC QLQ-C30 and EORTC QLQ-EN24; analysed with a repeated mixed model as one overall outcome over all time points
Worry including fear of recurrence | assessed at baseline, 6, 12, and 36 months after completion of primary treatment
  assessed with questionnaire: IOCv2; analysed with a repeated mixed model as one overall outcome over all time points
Worry including fear of recurrence | assessed at baseline, 6, 12, 36, and 60 months after completion of primary treatment
  assessed with questionnaire: IOCv2; analysed with a repeated mixed model as one overall outcome over all time points
Illness perceptions | assessed at baseline, 6, 12, and 36 months after completion of primary treatment
  assessed with questionnaire: BIPQ; analysed with a repeated mixed model as one overall outcome over all time points
Illness perceptions | assessed at baseline, 6, 12, 36, and 60 months after completion of primary treatment
  assessed with questionnaire: BIPQ; analysed with a repeated mixed model as one overall outcome over all time points
Anxiety and depression | assessed at baseline, 6, 12, and 36 months after completion of primary treatment
  assessed with questionnaire: HADS; analysed with a repeated mixed model as one overall outcome over all time points
Anxiety and depression | assessed at baseline, 6, 12, 36, and 60 months after completion of primary treatment
  assessed with questionnaire: HADS; analysed with a repeated mixed model as one overall outcome over all time points
Satisfaction with information provision | assessed at baseline, 6, 12, and 36 months after completion of primary treatment
  assessed with questionnaire: EORTC-INFO25; analysed with a repeated mixed model as one overall outcome over all time points
Satisfaction with information provision | assessed at baseline, 6, 12, 36, and 60 months after completion of primary treatment
  assessed with questionnaire: EORTC-INFO25; analysed with a repeated mixed model as one overall outcome over all time points
Health care providers' satisfaction with follow-up schedule (gynaecologist, (specialised) nurse) | assessed at 36 months after completion of primary treatment
  assessed with structured interviews/questionnaires
Health care providers' satisfaction with follow-up schedule (gynaecologist, (specialised) nurse) | assessed at 60 months after completion of primary treatment
  assessed with structured interviews/questionnaires
Time till recurrence | assessed at 36 months after completion of primary treatment
  In this study we will descriptively look at time till recurrence
Time till recurrence | assessed at 60 months after completion of primary treatment
  In this study we will descriptively look at time till recurrence
Survival | assessed at 36 months after completion of primary treatment
  descriptively look at survival
Survival | assessed at 60 months after completion of primary treatment
  descriptively look at survival

CONTACTS AND LOCATIONS:
Overall Officials: Lonneke van de Poll-Franse, PhD, Principal Investigator — Comprehensive Cancer Centre The Netherlands; Roy Kruitwagen, PhD, Principal Investigator — Maastricht University Medical Centre; Carien Creutzberg, PhD, Principal Investigator — Leiden University Medical Centre; Nicole Ezendam, PhD, Principal Investigator — Comprehensive Cancer Centre The Netherlands
Locations (47):
- Netherlands (47):
  - Jeroen Bosch, 's-Hertogenbosch
  - Noordwest ziekhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Amstelland Ziekenuis, Amstelveen
  - AMC, Amsterdam
  - AVL, Amsterdam
  - OLVG, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Bravis, Bergen op Zoom
  - Tergooi, Blaricum
  - Amphia, Breda
  - Reinier de Graaf Hospital, Delft
  - Deventer Hospital, Deventer
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Hospital, Eindhoven
  - Medical Spectrum Twente, Enschede
  - Groene Hart, Gouda
  - Martini Hospital, Groningen
  - UMC Groningen, Groningen
  - Röpcke-Zweers Ziekenhuis, Hardenberg
  - Tjongerschans, Heerenveen
  - Zuyderland Hospital, Heerlerheide
  - Westfries Gasthuis, Hoorn
  - Medical Center Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, Leiden
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - St. Antonius, Nieuwegein
  - Waterland Ziekenhuis, Purmerend
  - Bravis, Roosendaal
  - Franciscus Gasthuis, Rotterdam
  - Vlietland, Schiedam
  - Zuyderland, Sittard
  - Refaja, Stadskanaal
  - Haga hospital, The Hague
  - MC Haaglanden, The Hague
  - Elisabeth TweeSteden, TweeSteden, Tilburg
  - Elisabeth-TweeSteden, Tilburg
  - Bernhoven, Uden
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri, Venlo
  - Streekziekenhuis Koningin Beatrix, Winterswijk
  - Zuwe Hofpoort, Woerden
  - Zaans Medisch Centrum, Zaandam
  - Langeland, Zoetermeer
  - Gelre Ziekenhuizen, Zutphen
  - Isala kliniek, Zwolle

IPD SHARING:
Plan to Share IPD: No
After ending the study and analysis of the data, data becomes available for use by other researchers via PROFILES registry, according to the their terms

REFERENCES:
- [Derived] Ezendam NPM, de Rooij BH, Kruitwagen RFPM, Creutzberg CL, van Loon I, Boll D, Vos MC, van de Poll-Franse LV. ENdometrial cancer SURvivors' follow-up carE (ENSURE): Less is more? Evaluating patient satisfaction and cost-effectiveness of a reduced follow-up schedule: study protocol of a randomized controlled trial. Trials. 2018 Apr 16;19(1):227. doi: 10.1186/s13063-018-2611-x. PMID 29661218